CLINICAL TRIAL: NCT03180242
Title: Phase 1, Double-Blind, Randomized, Parallel-Group, Single-Dose, 3-Arm, Two-Stage, Comparative Pharmacokinetic Study of EirGenix' Trastuzumab and Herceptin® (Trastuzumab) Sourced From US and EU Administered to Healthy Male Volunteers
Brief Title: A Pharmacokinetic Study Comparing EG12014 and Herceptin (Trastuzumab) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EirGenix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EGC001
Record Dates: First submitted 2017-05-17; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- EG12014 (Experimental): EG12014
  Interventions: Biological: EG12014
- EU-sourced Herceptin (Active Comparator): EU-sourced Herceptin
  Interventions: Biological: EU-sourced Herceptin
- US-sourced Herceptin (Active Comparator): US-sourced Herceptin
  Interventions: Biological: US-sourced Herceptin

INTERVENTIONS:
Biological: EG12014 — EG12014, single-dose IV infusion over 90 min at 6 mg/kg
  Arms: EG12014
Biological: EU-sourced Herceptin — EU-sourced Herceptin, single-dose IV infusion over 90 min at 6 mg/kg
  Arms: EU-sourced Herceptin
Biological: US-sourced Herceptin — US-sourced Herceptin, single-dose IV infusion over 90 min at 6 mg/kg
  Arms: US-sourced Herceptin

SUMMARY:
The primary objective of this trial is to assess the pharmacokinetic similarity of EG12014 (Test IMP) compared to reference products sourced from the European Union (Reference IMP 1: Herceptin® 150 mg powder for concentrate for solution for infusion) and the United States (Reference IMP 2: Herceptin® 440 mg powder for concentrate for solution for infusion) after intravenous infusion over 90 minutes of a single dose of 6 mg/kg trastuzumab in 3 parallel groups of healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* male Caucasian subject
* age between 18 and 55 years (inclusive)
* physically and mentally healthy as judged by means of medical and standard laboratory examinations
* non-smokers or ex-smokers (stopped at least 6 months ago) with a smoking history of ≤5 pack-year equivalents (1 pack-year equivalent is equal to smoking 1 pack per day for 1 year ) and non-users of other nicotine containing products, confirmed by urine cotinine test
* BMI within the range (including the borders) of 18.5 to 30.0 kg/m2 and body weight not more than 105.0 kg
* Informed consent given in written form according to Section 5.4 of the protocol.

Exclusion Criteria:

* participation in another clinical trial at same time or within the preceding 3 months from the screening examination (calculated from the date of the final examination of the previous study)
* randomization into the present trial more than once
* blood donation or blood loss including plasmapheresis of >500 ml in the last 3 months before day 0 of the study
* history of drug abuse or use of illegal drugs: use of soft drugs, e.g. marihuana within 6 months of screening or hard drugs, e.g. cocaine, amphetamines, opioids, phencyclidine within 1 year of screening
* alcohol abuse, i.e. regular use of more than 2 units of alcohol per day or 10 units per week or a history of alcoholism (one unit of alcohol equals 250 ml beer, 125 ml wine or 25 ml spirits) or recovered alcoholics
* regular consumption of beverages or food containing methylxanthines (e.g. coffee, tea, cola, caffeine containing sodas, chocolate) equivalent to more than 500 mg methylxanthines per day
* positive drug screening and/or positive alcohol test at entry screening or on hospitalization day 0
* history of allergic diathesis or any clinically significant allergic disease (e.g. asthma or bronchial hyperreactivity, or allergic reactions to insect bites)
* any history of drug hypersensitivity (especially to the active and inactive ingredients of the trastuzumab preparation, or other monoclonal antibody or protein drugs) or intolerance to any sugar (e.g. fructose, glucose, or lactose)
* presence or a history of clinically significant cardiovascular, renal, hepatic, pulmonary, metabolic, endocrine, hematological, gastrointestinal, neurological, psychiatric or other diseases
* clinically significant illness within 4 weeks before day 0 of the study and during the study
* major surgery of the gastrointestinal tract except for appendectomy
* any chronic disease which might interfere with resorption, distribution, metabolism or excretion of the drug
* positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies
* administration of depot injectable solutions or medications with a half-life > 1 week (including study medications) within 6 months from day 0 of the study
* intake of enzyme-inducing, organotoxic or long half-life drugs, including prescription or OTC medications or herbal remedies (such as St. John's wort), within 4 weeks from day 0 of the study
* intake or administration of any systemic or topical medication within 2 weeks of day 0 of the study and during the study, except of up to a total dose of 1000 mg paracetamol or metamizole per day given in case of an adverse event (e.g. IRR's: pyrexia, headache) during the study
* intake of drugs known to alter the major organs or systems such as barbiturates, phenothiazines, cimetidine, omeprazole etc. within the last 2 months
* previous exposure to a monoclonal antibody drug or current or expected use of other biological products.
* systolic blood pressure outside the range of 100 to 140 mmHg and/or diastolic blood pressure outside the range of 60 to 90 mmHg at screening and on day 0
* heart rate outside the range of 50 to 90 beats/min at screening and on day 0
* axillary body temperature outside the interval of 35.5 to 37.1°C at screening and on day 0
* any clinically significant abnormality of the resting ECG (12-lead) (i.e. AV block, 2° to 3°, sinus bradycardia, sick sinus syndrome, SA block)
* laboratory values outside normal range with clinical relevance at screening examination and on day 0 of the study
* special diet due to any reason, e.g. vegetarians
* not fulfilling study specific restrictions given in Sections 9.4 Restrictions and 9.6 Diet of the protocol
* any planned surgery within 78 days after dosing on day 1
* subjects who are known or suspected: not to comply with the study directives or meet the required visit schedules; not to be reliable or trustworthy; not to be capable of understanding and evaluating the information given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed; to be in such a precarious financial situation that they no longer weigh up the possible risks of their participation and the unpleasantness they may be involved in.
* left ventricular ejection fraction (LVEF) <55%, assessed by means of transthoracic echocardiography .

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2016-08-22 (Actual); Study Completion 2016-08-22 (Actual)

PRIMARY OUTCOMES:
Area under the concentration/time curve, from time 0 h extrapolated to infinity (AUC(0-∞)) | 70 days

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 70 days
Area under the concentration/time curve, calculated by the trapezoidal rule from time 0 h to last observed concentration at time t (AUC(0-t)) | 70 days
Residual area in percent (AUCres) | 70 days
Serum concentration half-life (t½) | 70 days
Adverse events | 70 days
Clinical laboratory values | 70 days
Local tolerability at infusion site | 70 days
Vital signs and physical examination results | 70 days
Electrocardiogram (ECG) measurements | 70 days
Incidence of anti-drug antibodies (ADA) | 70 days